CLINICAL TRIAL: NCT03448601
Title: Specialized Centers of Excellence for Research on Minority Health and Health Disparities: Alzheimer's Disease and Precision Medicine Research: Addressing Gaps in Participation of American Indian and Alaska Native People
Brief Title: Alzheimer's Disease and Precision Medicine Research Among Native People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Washington State University (Other); Missouri Breaks Industries Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-1627
Record Dates: First submitted 2018-02-09; First posted 2018-02-28 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
Keywords: Precision Medicine
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in equal proportions either to receive 1) a standard, non-tailored educational brochure on Alzheimer's Disease (AD), the value of precision medicine (PM), and the importance of research (control); OR 2) to receive a culturally tailored brochure with graphics and identical information; OR 3) to view a digital story featuring personal narratives of AI/ANs (intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-tailored control group (No Intervention): Participates will read the standard Alzheimer's disease and Precision Medicine brochure with standard text-based content NOT specifically tailored for AI/ANs.
- Culturally tailored video intervention group (Experimental): Participants will view a short 5-minute culturally-tailored video.
  Interventions: Other: Culturally tailored video intervention group
- Culturally tailored brochure intervention group (Experimental): Participants will read a culturally-tailored educational brochure on Alzheimer's disease and Precision Medicine.
  Interventions: Other: Culturally tailored brochure intervention group

INTERVENTIONS:
Other: Culturally tailored brochure intervention group — Culturally-tailored Alzheimer's Disease and precision medicine educational brochure.
  Arms: Culturally tailored brochure intervention group
Other: Culturally tailored video intervention group — Culturally-tailored Alzheimer's Disease and precision medicine educational video.
  Arms: Culturally tailored video intervention group

SUMMARY:
This project intends to address the gaps in Alzheimer's disease (AD) and precision medicine (PM) research in American Indian and Alaska Native (AI/AN) populations by comparing written and video-based materials for recruitment into AD and PM research, and by creating an AD-PM registry of AI/AN individuals who are willing to be contacted for future research opportunities.

DETAILED DESCRIPTION:
This project intends to address the gaps in Alzheimer's disease (AD) and precision medicine (PM) research in American Indian and Alaska Native (AI/AN) populations by comparing written and video-based materials for recruitment into AD and PM research, and by creating an AD-PM registry of AI/AN individuals who are willing to be contacted for future research opportunities. The project will be a 3-arm RCT with a sample size of 501 AI/AN adults, aged 40 years and older. The RCT enables us to compare outcomes between groups to determine the effect of a tailored brochure and video compared to non-tailored, text-based recruitment materials, and assemble a large registry of AI/ANs with biospecimens and data from medical records for future AD research.

The AI/AN population is growing as a proportion of the total US population, and gains in life expectancy mean that the number of Native elders at risk of AD is rapidly increasing. Therefore, there is a need for research in this understudied group.

The study procedures are expected to take participants approximately 2-3 hours to finish. Participants will be asked to complete a pre-intervention self-report questionnaire and have their height, weight, and neck circumference measured. Next, they will be randomized to one of the 3-treatment arms. Participants allocated to the control condition will receive the standard brochure on AD and PM, with standard text-based content not specifically tailored for AI/ANs. Participants randomized to the intervention will either view a short culturally tailored video (5 minutes) or read a culturally tailored educational brochure. All brochures and video will contain the same base information on AD and PM. Participants will have as much time as they need to review the material. After each participant has finished reading the relevant brochure or viewing the video, they will be asked to complete post-intervention data collection that includes: 1) an ADRD knowledge questionnaire and 2) enrollment in the AD-PM Registry. If the participant chooses not to enroll in the AD-PM Registry, their participation in the study is complete. If the participant agrees to enroll in the registry, they will be asked to complete 3) the AD-PM Module, 4) biospecimen donation (blood, saliva, and urine samples), and 5) permission to access medical records. Participants who complete the AD-PM module and provide biospecimens but decline consent to access medical records will still be added to the registry.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as American Indian or Alaska Native
* able to speak, read, and understand English
* age 40 or older
* has cognitive and decisional capacity to consent

Exclusion Criteria:

* do not speak or read English
* vision or hearing impairments that would prevent reading a brochure or watching a video

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
AD-PM Module Completion | Baseline
  Completion of the AD-PM Module will be assessed by binary (yes, no) indicators of 1) providing consent for the Module; and 2) answering a question about enrolling in the AD-PM cohort and by a variable summarizing the total number of missing responses for the AD-PM module questions.
Cohort Enrollment Questionnaire | Baseline
  Enrollment in the AD-PM Cohort will be assessed by binary (yes, no) indicators of agreeing to 1) join the Cohort, and 2) be contacted for participation in future studies.

SECONDARY OUTCOMES:
Willingness to Participate in Research Questionnaire | Baseline
  Willingness to participate will be rated using a 4-point Likert scale (1=definitely would not, 2=probably would not; 3=probably would; 4=definitely would) after viewing 4 vignettes portraying hypothetical future projects related to Alzheimer's Disease, dementia, and Precision Medicine. Ranges for each vignette are 1 to 4 with higher scores indicating greater willingness to participate in research.
Alzheimer's Disease (AD) Knowledge Scale | Baseline
  30 true/false items on risk factors, assessment, diagnosis, symptoms, life impact, caregiving, treatment, and management. Range is 0 - 30 with higher scores indicating greater AD knowledge.
Attitudes about Precision Medicine self-report survey | Baseline
  Investigators will adapt a 44-item survey created by the National Institutes of Health to measure attitudes about the "All of Us" Alzheimer's Disease/Precision Medicine (AD/PM) Research Program to approximately 20 items specifically related to attitudes about PM rather than on All of Us more broadly. Items will be multiple choice (Definitely yes, Probably yes, Probably no, Definitely no) and binary (agree, disagree; yes, no). Ranges are not yet established as the survey is under development. Higher scores will indicate more positive attitudes about PM.
Self-Administered Gerocognitive Exam (SAGE) | Baseline
  To measure baseline cognitive function, scores from SAGE ranging from normal to mild cognitive impairment. Test scores range from 22 (normal) to 15 (mild cognitive impairment), with a score < 14 indicative of dementia and a score of ≥ 17 considered normal.
Orthogonal Cultural Identification Scale | Baseline
  Cultural identity will be assessed from ratings of the degree to which participants identify with Native and White ways of life in family and community interactions. Items range from 1=not at all, 2=not much, 3=some, to 4=a lot with higher scores indicating higher cultural identification with the culture described.

CONTACTS AND LOCATIONS:
Overall Officials: Spero Manson, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Missouri Breaks Industries Research, Inc., Rapid City, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta KM, Yaffe K, Perez-Stable EJ, Stewart A, Barnes D, Kurland BF, Miller BL. Race/ethnic differences in AD survival in US Alzheimer's Disease Centers. Neurology. 2008 Apr 1;70(14):1163-70. doi: 10.1212/01.wnl.0000285287.99923.3c. Epub 2007 Nov 14. PMID 18003939
- [Background] Castor ML, Smyser MS, Taualii MM, Park AN, Lawson SA, Forquera RA. A nationwide population-based study identifying health disparities between American Indians/Alaska Natives and the general populations living in select urban counties. Am J Public Health. 2006 Aug;96(8):1478-84. doi: 10.2105/AJPH.2004.053942. Epub 2006 Mar 29. PMID 16571711